CLINICAL TRIAL: NCT01130415
Title: Is the Method of Screening in Sacral Neuromodulation a Prognostic Factor for Long-term Success?
Brief Title: Screening Method in Sacral Neuromodulation
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Scientific Foundation Urology Maastricht (Unknown)
Responsible Party: P. van Kerrebroeck, Maastricht University Medical Centre
Other Study IDs: 1234
Record Dates: First submitted 2010-05-19; First posted 2010-05-26 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Overactive Bladder; Urinary Retention
Keywords: Sacral neuromodulation; Screening; Percutaneous nerve evaluation; Tined lead
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with sacral neuromodulation

SUMMARY:
The purpose of this study was to evaluate whether there is a difference in long-term outcome between patients screened with the percutaneous nerve evaluation (PNE) and first stage tined lead procedure (TLP).

DETAILED DESCRIPTION:
Purpose: To evaluate if there is a difference in long-term outcome of sacral neuromodulation (SNM) between patients screened with the percutaneous nerve evaluation (PNE) and first stage tined lead procedure (TLP). Furthermore, we wanted to evaluate the outcome in patients who only responded to screening with TLP after failure of initial PNE.

Materials and methods: We evaluated all patients screened for eligibility to receive SNM treatment since the introduction of the tined lead technique in our centre in 2002. In May 2009, all implanted patients were asked to keep a voiding diary to record the effect of SNM on urinary symptoms. Success was defined as more than 50% improvement in at least one of the relevant voiding diary parameters compared to baseline. Chi square analysis was used to evaluate differences in long-term outcome for the separate screening methods.

Results: In total, 92 patients were screened for SNM. Of the 76 patients who were screened with PNE, 35 (46%) met the criteria for permanent implantation, whereas 11 of the 16 patients (69%) who underwent direct screening with TLP had permanent stimulators placed. Of the 41 patients who failed PNE and subsequently underwent screening with TLP, 18 (44%) were implanted with an INS after showing a successful response. The mean follow-up was 53 months (range 35-77 months) at the time of voiding diary analysis. Statistical analysis showed no difference between type of screening and long-term success (p=0.94).

Conclusion: Although first stage TLP is a more reliable screening tool than PNE, the long-term success rate does not seem to be dependent on the screening method. Furthermore, patients who initially failed PNE but responded to prolonged screening with TLP, appear to be at least as successful in the long-term as patients who directly responded to PNE or TLP.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been treated for overactive bladder syndrome or chronic non-obstructive urinary retention with sacral neuromodulation by using the tined lead

Exclusion Criteria:

* patients with bilateral implantation of a tined lead
* patients who have been treated with sacral neuromodulation for pelvic pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been treated with sacral neuromodulation in our centre between 2002 and 2009
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2002-05; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
long-term success measured with voiding diaries | 5 years
  Successful treatment was defined as more than 50 percent improvement in the key voiding diary variables compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Philip van Kerrebroeck, Prof, Study Director — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands